CLINICAL TRIAL: NCT02659293
Title: Phase 3 Randomized Trial of Carfilzomib, Lenalidomide, Dexamethasone Versus Lenalidomide Alone After Stem-cell Transplant for Multiple Myeloma
Brief Title: Trial of Carfilzomib, Lenalidomide, Dexamethasone Versus Lenalidomide Alone After Stem-cell Transplant for Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1286
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; stem-cell transplant; Symptomatic myeloma; lenalidomide; carfilzomib; dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Control) (Active Comparator): Treatment with lenalidomide only
  Interventions: Drug: Lenalidomide (Control)
- Experimental Combination Regimen (Experimental): Experimental arm using a combination of Carfilzomib, Lenalidomide and Dexamethasone
  Interventions: Drug: Lenalidomide; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — * Cycle 1: 15 mg days 1-21
  * Cycles 2-4: 25 mg days 1-21 if tolerated, otherwise continue at lower dose
  * Cycles 5 and beyond: best tolerated dose days 1-21
  Other Names: Revlimid
  Arms: Experimental Combination Regimen
Drug: Carfilzomib — * Cycle 1: 20 mg/m2 Days 1, 2; 36 mg/m2 Days 8, 9, 15, 16. Alternatively, intermediate dose escalation (to 27mg/m2 on days 8,9 of cycle 1) will be al12,lowed at the treating physician's discretion.
  * Cycle 2-4: 36 mg/m2 if tolerated Days 1, 2, 8, 9, 15, 16
  * Cycles 5-8 (patients that are MRD- and have no risk factors at the end of cycle 6) and Cycle 5 - 36 (for MRD+ patients and high risk patients at the end of cycle 6): best tolerated dose Days 1, 2, 15, 16
  Other Names: Kyprolis
  Arms: Experimental Combination Regimen
Drug: Dexamethasone — * Cycles 1 - 4: 20 mg PO or IV per dose Days 1, 8, 15, 22
  * Cycles 5+: 20 mg or best tolerated dose PO or IV per dose Days 1, 8, 15, 22
  Arms: Experimental Combination Regimen
Drug: Lenalidomide (Control) — * Cycles 1-4: Days 1-28. Lenalidomide will begin at a dose of 10 mg PO daily (2 capsules per day). After three months, the dose will be increased, provided ANC ≥ 1,000/µL, platelet count ≥ 75,000/µL, and all nonhematologic toxicity is ≤ grade 1, to 15 mg PO daily (3 capsules per day).
  * Cycles 5 and beyond: best tolerated dose days 1-28
  Other Names: Revlimid
  Arms: Lenalidomide (Control)

SUMMARY:
This is a Phase 3 randomized trial of carfilzomib, lenalidomide, dexamethasone versus lenalidomide alone after stem-cell transplant for multiple myeloma, eligible to subjects who completed autologous stem cell transplant for symptomatic myeloma who are considered for lenalidomide maintenance.

DETAILED DESCRIPTION:
Primary Objective:

* To compare progression free survival between Kyprolis (Carfilzomib), Revlimid (lenalidomide), Dexamethasone (KRd) arm and lenalidomide arm

Secondary Objectives

* To determine the rate of minimal residual negative disease (MRD) at 6 and 12 months after randomization
* To compare the efficacy (rate of partial response, very good partial response, complete response, and stringent complete response) of KRd vs. Lenalidomide alone after randomization

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed single autologous stem cell transplant after completion of at most 2 induction regimens (excluding dexamethasone alone) and are in at least stable disease in the first 100 days after stem cell transplantation.
2. Patients must be within 12 months of initiation of induction therapy and must have had not more than 2 prior induction regimens.
3. Bone marrow specimen will be required at study entry; available DNA sample will be used for calibration step for MRD evaluation by gene sequencing.
4. Males and females ≥ 18 years of age
5. ECOG performance status of 0-1
6. Adequate hepatic function, with bilirubin ≤ 1.5 x ULN and aspirate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN
7. ANC ≥ 1.0 x 109/L, hemoglobin ≥ 8 g/dL, platelet count ≥ 75 x 109/L.
8. Calculated creatinine clearance (by Cockcroft-Gault) ≥ 50 ml/min or serum creatinine below 2 mg/dL
9. Females of childbearing potential (FCBP) must have 2 negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to initiating lenalidomide. The first pregnancy test must be performed within 10-14 days before and the second pregnancy test must be performed within 24 hours before lenalidomide is prescribed for Cycle 1 (prescriptions must be filled within 7 days).
10. FCBP must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting lenalidomide; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study.

    UCM IRB CRd vs. R Version 1.0 Page 11
11. Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
12. All study participants in the US must be consented to and registered into the mandatory Revlimid REMS® program and be willing and able to comply with the requirements of Revlimid REMS®.
13. Voluntary written informed consent

Exclusion Criteria:

1. Patients who have had more than 12 months of prior therapy. Patients outside of this window may be considered for inclusion on a case-by-case basis.
2. Patients who progressed after initial therapy.

   1. Subjects whose therapy changed due to suboptimal response, intolerance, etc., remain eligible, provided they do not meet criteria for progression.
   2. No more than two regimens for induction will be allowed excluding dexamethasone alone.
3. Evidence of progressive disease as per International Myeloma Working Group (IMWG) criteria
4. Patients who have already started or received post-transplant maintenance or consolidation regimen
5. Patients not able to tolerate lenalidomide or carfilzomib or dexamethasone
6. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
7. Plasma cell leukemia
8. Waldenström's macroglobulinemia or IgM myeloma
9. Peripheral neuropathy ≥ Grade 2 at screening
10. Diarrhea > Grade 1 in the absence of antidiarrheals
11. CNS involvement
12. Pregnant or lactating females
13. Radiotherapy within 14 days before randomization. Seven days may be considered if to single area.
14. Major surgery within 3 weeks prior to first dose
15. Myocardial infarction within 6 months prior to enrollment, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
16. Prior or concurrent deep vein thrombosis or pulmonary embolism
17. Rate-corrected QT interval of electrocardiograph (QTc) > 470 msec on a 12-lead ECG during screening
18. Uncontrolled hypertension or diabetes
19. Acute infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
20. Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
21. Non-hematologic malignancy or non-myeloma hematologic malignancy within the past 3 years except a) adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, or prostate cancer < Gleason Grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone
22. Any clinically significant medical disease or condition that, in the Treating Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rates in participants receiving drug combination | 4 years
  Measurement of time to disease worsening as measured by International Myeloma Working Group (IMWG) response criteria.

SECONDARY OUTCOMES:
Rate of minimal residual negative disease (MRD) in participants receiving drug combination | 3 years
  Calculation of number of participants with MRD-negative disease.
Response rate in participants receiving drug combination | 3 years
  Number of participants with disease response (e.g. improvement) as measured by International Myeloma Working Group (IMWG) response criteria.
Treatment-related side effects | From date of screening until end of treatment
  Number of participants with grade 2 or greater treatment-related side effects as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Jakubowiak, MD, PhD, Principal Investigator — University of Chicago
Locations (3):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Wayne State University - Karmanos Cacner Institute, Detroit, Michigan
- Polish Myeloma Consortium, Poznan, Poland

REFERENCES:
- [Derived] Kubicki T, Jamroziak K, Robak P, Czyz J, Tyczynska A, Druzd-Sitek A, Giannopoulos K, Wrobel T, Nowicki A, Szczepaniak T, Lojko-Dankowska A, Matuszak M, Gil L, Pula B, Szukalski L, Konska A, Zaucha JM, Walewski J, Mikulski D, Czabak O, Robak T, Kruk-Kwapisz D, Derman BA, Major A, Jakubowiak AJ, Dytfeld D. Health-related quality of life in patients with multiple myeloma treated in the phase 3 ATLAS trial of post-transplant maintenance with carfilzomib, lenalidomide, and dexamethasone or lenalidomide alone. Pol Arch Intern Med. 2024 May 28;134(5):16749. doi: 10.20452/pamw.16749. Epub 2024 May 14. No abstract available. PMID 38747414
- [Derived] Kubicki T, Dytfeld D, Barnidge D, Sakrikar D, Przybylowicz-Chalecka A, Jamroziak K, Robak P, Czyz J, Tyczynska A, Druzd-Sitek A, Giannopoulos K, Wrobel T, Nowicki A, Szczepaniak T, Lojko-Dankowska A, Matuszak M, Gil L, Pula B, Szukalski L, Konska A, Zaucha JM, Walewski J, Mikulski D, Czabak O, Robak T, Jiang K, Cooperrider JH, Jakubowiak AJ, Derman BA. Mass spectrometry-based assessment of M protein in peripheral blood during maintenance therapy in multiple myeloma. Blood. 2024 Aug 29;144(9):955-963. doi: 10.1182/blood.2024024041. PMID 38713888
- [Derived] Dytfeld D, Wrobel T, Jamroziak K, Kubicki T, Robak P, Walter-Croneck A, Czyz J, Tyczynska A, Druzd-Sitek A, Giannopoulos K, Nowicki A, Szczepaniak T, Lojko-Dankowska A, Matuszak M, Gil L, Pula B, Rybka J, Majcherek M, Usnarska-Zubkiewicz L, Szukalski L, Konska A, Zaucha JM, Walewski J, Mikulski D, Czabak O, Robak T, Lahoud OB, Zonder JA, Griffith K, Stefka A, Major A, Derman BA, Jakubowiak AJ. Carfilzomib, lenalidomide, and dexamethasone or lenalidomide alone as maintenance therapy after autologous stem-cell transplantation in patients with multiple myeloma (ATLAS): interim analysis of a randomised, open-label, phase 3 trial. Lancet Oncol. 2023 Feb;24(2):139-150. doi: 10.1016/S1470-2045(22)00738-0. Epub 2023 Jan 12. PMID 36642080